CLINICAL TRIAL: NCT05960136
Title: The Impact of COVID-19 on the Rate of Peri-operative Complications of Maxillary Sinus Floor Augmentation Procedure.
Brief Title: Impact of COVID-19 on Sinus Augmentation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Kadry, Lecturer of oral and Maxillofacial Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-19 and sinus lift
Record Dates: First submitted 2023-07-22; First posted 2023-07-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinus lift in patients with previous COVID-19 infection (Active Comparator): Sinus floor augmentation in the posterior atrophic maxilla with delayed implant placement in patients with positive history of previous COVID-19 infection.
  Interventions: Procedure: Sinus lift in patients with positive COVID-19 history
- Sinus lift in patients with negative history of previous COVID (Active Comparator): Sinus floor augmentation in the posterior atrophic maxilla with delayed implant placement in patients with negative history of COVID-19 infection.
  Interventions: Procedure: Sinus lift with negative COVID-19 history

INTERVENTIONS:
Procedure: Sinus lift in patients with positive COVID-19 history — Sinus augmentation in the posterior atrophic maxilla in patients with positive COVID-19 history
  Arms: Sinus lift in patients with previous COVID-19 infection
Procedure: Sinus lift with negative COVID-19 history — Sinus augmentation in the posterior atrophic maxilla in patients with negative COVID-19 history
  Arms: Sinus lift in patients with negative history of previous COVID

SUMMARY:
The risk of Schneiderian membrane perforation and the postoperative complications of the sinus floor elevation surgery were evaluated for patients with and without history of COVID-19 infection.

DETAILED DESCRIPTION:
COVID-19 induced chronic sinusitis with subsequent increased Schneiderian membrane thickness could increase the risk of its perforation during the sinus floor elevation. The aim of the study is to compare the incidence of Schneiderian membrane perforation and the postoperive complications of the sinus floor elevation in patients with and without history of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 4 mm or less residual alveolar bone height
* Age more than 18 years
* Highly motivated patients

Exclusion Criteria:

* Patients who suffer from any systemic disease
* sinus pathosis other than sinusitis induced covid 19
* Patients under any medication that may interfere with the normal bone healing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Sinus membrane perforation | Duration sinus lift
  Intraoperative assessment of the incidence of sinus membrane perforation

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Awadallah, Study Chair — Lecturer at Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt